CLINICAL TRIAL: NCT06139926
Title: Clinical Study of Dexmedetomidine Administered Intranasally to Relieve Perioperative Anxiety and Depression in Patients With Colorectal Tumors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Sixu Lai, cinical investigator, First Affiliated Hospital of Chongqing Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023328
Record Dates: First submitted 2023-11-15; First posted 2023-11-18 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine administered intravenously (Other): Dexmedetomidine was administered intravenously 15 min prior to patient induction (concentration 4 μg/ml; loading dose 1 μg/kg for 15 min; maintenance dose: 0.2 μg/(kg.h) until surgical specimen removal).
  Interventions: Drug: Dexmedetomidine administered intranasally
- Dexmedetomidine administered intranasally (Experimental): Intranasal administration of dexmedetomidine (original solution) was given at the bedside of the ward as per the pre-tested recommended dose. The patient's vital signs were maintained. On the day of surgery, 30 min before induction of anesthesia, intranasal dexmedetomidine (original solution) was administered in the operating room at the pre-tested recommended dose.
  Interventions: Drug: Dexmedetomidine administered intranasally

INTERVENTIONS:
Drug: Dexmedetomidine administered intranasally — Intranasal administration of dexmedetomidine (plain) was given at the bedside of the ward as per the pre-tested recommended dose. The patient's vital signs were maintained. On the day of surgery, 30 min before induction of anesthesia, intranasal dexmedetomidine (original solution) was administered in the operating room at the pre-tested recommended dose.

SUMMARY:
Currently, domestic and international research on dexmedetomidine as well as anxiety and depression is more focused on basic research. In terms of clinical research, dexmedetomidine is more often used in pediatrics, short surgeries, intensive care units, etc., for sedation and analgesia; while less research has been done for the relief of anxiety and depression. At present, on the one hand, the number of oncology patients is on the rise both at home and abroad, and on the other hand, anxiety and depression account for an increasing proportion of healthcare in the world. Tumor patients, as a high prevalence group of anxiety and depression, their prognosis and regression are also more complicated. Therefore, exploring the role of intranasal administration of dexmedetomidine in relieving perioperative anxiety and depression in oncology patients has a very strong practical basis and clinical significance.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a preoperative diagnosis of colorectal cancer who were to undergo their first oncologic procedure
2. Patients who opted for general anesthesia via orotracheal intubation
3. Age ≥18 years old
4. ASA classification II-III (5) 18.0 < BMI < 30.0
5. Signed informed consent.

Exclusion Criteria:

1. Diagnosed mental illness or cognitive impairment, or taking antipsychotic, sedative-hypnotic, or anxiolytic-depressant medications
2. Serious abnormalities of liver or kidney function.
3. Prior alcohol or drug abuse
4. Second or third degree atrioventricular block, severe sinus bradycardia (<50 beats/min), sick sinus node syndrome, congenital heart disease, and other cardiac arrhythmias that severely affect hemodynamic stability
5. Grade 3 hypertension
6. Any disease of the head, such as cerebral infarcts, epilepsy, head trauma, etc.
7. Confirmed diagnosis of non-tumor-induced chronic ( ≥3 months) neuropathic pain
8. Inability to understand the meaning of the scale and complete the scoring.
9. Women preparing for pregnancy, pregnant women, or breastfeeding
10. Patients with myasthenia gravis
11. Respiratory function score ≥3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes in perioperative HADS scale scores. | The first HADS scale score was performed at preoperative follow-up, and multiple HADS scale scores were performed within 30 days of surgery to observe changes in scores
  The first HADS scale score was performed at preoperative follow-up, and multiple HADS scale scores were performed within 30 days of surgery to observe changes in scores.The scale has a minimum score of 0 and a maximum score of 21. Higher scores indicate greater levels of anxiety or depression.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China